CLINICAL TRIAL: NCT05841979
Title: The Lived Experiences Measured Using Rings Pilot Study
Acronym: LEMURS-P
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: MassMutual - Private Industry Funded (Unknown)
Responsible Party: Principal Investigator, Matthew Price, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEMURS S23
Record Dates: First submitted 2023-04-06; First posted 2023-05-03 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-03

CONDITIONS: Depression; Stress; Sleep; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- group-based therapy (Experimental): Group therapy delivered via moodlifters
  Interventions: Behavioral: Moodlifters
- physical activity (Experimental): Physical Activity and Exercise
  Interventions: Behavioral: Physical Activity
- nature experience (Experimental): Nature Experiences
  Interventions: Behavioral: Nature Experiences
- self-monitoring (No Intervention): Placebo control

INTERVENTIONS:
Behavioral: Moodlifters — Mood Lifters, a novel mental wellness program, was developed as a more accessible means to provide psychotherapy (Votta & Deldin, 2022). Meetings covered biopsychosocial areas and skills that were drawn from multiple therapeutic interventions consistent with a biopsychosocial framework. Areas included physical health, negative thoughts, problem-solving, emotional awareness and regulation, building relationships, behavioral activation, and using a strengths-based approach. ML is delivered by peer leaders who are individuals that have completed the program as well as a training program.
  Arms: group-based therapy
Behavioral: Physical Activity — Participants randomized to the exercise arm received 14 weeks of a structured weekly strength and conditioning training program to enhance muscle mass, strength, cardiorespiratory fitness, and overall well-being. The program is based on previous research showing that cardiorespiratory fitness and muscle strength/size can both contribute to decreased mortality/increased longevity and enhanced mental health (Burke et al., 2017; McLeod et al., 2016; Srikanthan & Karlamangla, 2014; Strasser & Burtscher, 2018). The training program consists of three training sessions per week, with one being an in-person group session guided by a certified strength and conditioning specialist. The other two training sessions are self-guided via the mobile app Trainheroic. This weekly training schedule aligns with previous research showing benefits to structuring an exercise program using a variety of social contexts (group setting, own, etc.; Burke et al., 2017).
  Arms: physical activity
Behavioral: Nature Experiences — Participants randomized to the Nature Experiences participated in 14 weeks of group and self-directed activities to connect with the natural environment. Weekly group activities will be led by Nature Guides, who are undergraduate and graduate students with extensive outdoor education training. Group activities will last one hour a week and include hiking in forests, walking in parks, bird-watching, mindfulness exercises, and snow activities. Participants will be given a list of self-directed activity suggestions each week. The goal of self-directed activities is to spend an additional two hours in a natural environment each week.
  Arms: nature experience

SUMMARY:
The transition to college is a period of elevated risk for a range of mental health conditions. For students with pre-existing mental health diagnoses, the added pressures can exacerbate challenges. Although colleges and universities strive to provide mental health support to their students, the high demand for these services makes it difficult to provide scalable cost-effective solutions. To address these issues, the present study aims to compare the efficacy of three different treatments using a large cohort of 600 students transitioning to college. Interventions were selected based on their potential for generalizability and cost-effectiveness on college campuses. The randomized controlled trial will assign 150 participants to one of four arms: 1) group-based therapy, 2) physical activity program, 3) nature experiences group, or 4) self-monitoring condition as the control group. In addition, biometric data will be collected from all participants using a wearable device to develop algorithmic predictions of mental and physical health functioning. Once recruitment is complete, modeling strategies will be used to evaluate the outcomes and effectiveness of each intervention. The findings of this study will provide evidence as to the benefits of implementing scalable and proactive interventions using technology with the goal of improving well-being and success of new college students.

ELIGIBILITY:
Inclusion Criteria:

* Current undergraduate student in their first year of school
* own a mobile device

Exclusion Criteria:

* None

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Depression as measured by Depression, Anxiety, Stress Survey - 21 (Depression subscale) | Change in depression scores from time of randomization through 5 months
  Self Reported Depression
Anxiety as measured by Depression, Anxiety, Stress Survey - 21 (Anxiety subscale) | Change in anxiety scores from time of randomization through 5 months
  Self ReportedAnxiety
Stress as measured by Depression, Anxiety, Stress Survey - 21 (Stress subscale) | Change in stress scores from time of randomization through 5 months
  Self Reported Stress
Well-Being as measured by Warwick-Edinburgh Mental Well-being Scale | Change in well-being scores from time of randomization through 5 months
  Self Reported well-being
Stress as measured by the Perceived Stress Scale | Change in stress scores from time of randomization through 5 months
  Self Reported subclinical stress

SECONDARY OUTCOMES:
Sleep Quality Index | Change in sleep quality scores from time of randomization through 5 months
  Self Reported Sleep
Oura Ring Sleep Index | Change in Oura Sleep measured scores from time of randomization through 5 months
  Biometric Sleep recorded from an Oura Ring
Medical Outcomes Social Support Survey | Change in social support scores scores from time of randomization through 5 months
  Social Support

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bloomfield, MD, PhD, Principal Investigator — University of Vermont; Chris Danforth, PhD, Principal Investigator — University of Vermont; Ryan McGinnis, PhD, Principal Investigator — University of Vermont; Ellen McGinnis, PhD, Principal Investigator — University of Vermont; Matthew Price, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Price M, Hidalgo JE, Bird YM, Bloomfield LSP, Buck C, Cerutti J, Dodds PS, Fudolig MI, Gehman R, Hickok M, Kim J, Llorin J, Lovato J, McGinnis EW, McGinnis RS, Norton R, Ramirez V, Stanton K, Ricketts TH, Danforth CM. A large clinical trial to improve well-being during the transition to college using wearables: The lived experiences measured using rings study. Contemp Clin Trials. 2023 Oct;133:107338. doi: 10.1016/j.cct.2023.107338. Epub 2023 Sep 16. PMID 37722484